CLINICAL TRIAL: NCT01565031
Title: A Simple Prognostic Score for Future Risk Assessment in Patients With Controlled Asthma Who Undergo a Step-down Guidelines-based Strategy
Brief Title: Prediction of Future Risk in Patients With Controlled Asthma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Luis Perez de Llano (Other)
Collaborators: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other); Hospital Clinic of Barcelona (Other); Hospital Galdakao-Usansolo (Other Government); Complexo Hospitalario Universitario de A Coruña (Other)
Responsible Party: Sponsor-Investigator, Luis Perez de Llano, MD, PhD., Hospital Universitario Lucus Augusti
Organization: Hospital Universitario Lucus Augusti (Other)
Other Study IDs: HULA
Record Dates: First submitted 2012-03-26; First posted 2012-03-28 (Estimated); Last update posted 2012-03-28 (Estimated); Status verified 2012-03

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- controlled asthmatics, down-titration: Adults (age between 18 and 80) with asthma under control (see definitions) during the last 3 months, treated with a combination of ICS and long-acting beta-agonist (LABA).
  Interventions: Procedure: Step-wise down-titration according to international guidelines.

INTERVENTIONS:
Procedure: Step-wise down-titration according to international guidelines. — The medication will be adjusted according to each patient´s level of control. Depending on the state of control of asthma, the dose will be adjusted up or down (step-up therapy and step-down therapy, respectively) in accordance with GINA.

SUMMARY:
The optimal score to predict unfavourable outcome in well-controlled asthma patients who are undergoing a step-wise down-titration of their medication is still lacking. Thus, a study is warranted to prospectively develop a prognostic system -easy to perform (suitable for use in the clinical rather the research setting)- for asthmatic patients in this clinical setting.

HYPOTHESIS: A simple score system can accurately predict clinical deterioration of asthma in well-controlled patients who are undergoing a step-wise down-titration of their medication according to international guidelines.

METHODS The investigators designed a prospective, multicenter, observational study at five centers in cities across Spain.

The patients group (N = 225) will be evaluated to produce a clinical prediction rule for loss of control. The investigators will consider the following variables in the risk factor analysis: documented history of previous bronchial obstruction (FEV1/FVC < 70%), coefficient of variation (CV) of morning peak expiratory flow (PEF), history of exacerbations, fraction of exhaled nitric oxide (FENO), Asthma control test (ACT), ACT item 3 and adherence.

The score model will be prospectively validated in an independent set of 113 patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age between 18 and 80.
* Asthma under control during the last 3 months.
* Treated with a combination of ICS and long-acting beta-agonist (LABA.
* Classified as "moderate asthma" by their attending physician.

Exclusion Criteria:

* Active smoking.
* Pregnancy.
* Treatment with oral corticosteroids, omalizumab or immunotherapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Well-controlled asthmatics who are regularly under the care of Allergy or Pneumology specialists.
Sampling Method: Non-Probability Sample
Enrollment: 338 (Estimated)
Dates: Start 2012-05; Primary Completion 2015-05 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Loss of asthma control. | 12 months
  Loss of control: Either ACT score ≤ 19 or the development of exacerbation or FEV1 decrease ≥20%.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Perez de Llano, Md, PhD, Principal Investigator — Servicio Galego de Saude
Locations (1):
- Pneumology Service, Lugo, Lugo, Spain